CLINICAL TRIAL: NCT07086872
Title: Impact of Adding Integrated Neuromuscular Inhibition Technique to Mulligan Therapy in Symptomatic Forward Head Posture
Acronym: FHP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Al Shaymaa Shaaban Abd El Azeim, principle investigator : alshaymaa shaaban abd el azeim, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005806
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Forward Head Posture
Keywords: Integrated Neuromuscular Inhibition Technique; Mulligan Therapy; Forward Head Posture

STUDY DESIGN:
Intervention Model Description: integrated neuromuscular inhibition and mulligan
Who Masked: Outcomes Assessor
Masking Description: opaque sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Integrated Neuromuscular Inhibition Technique and mulligan therapy (Experimental): thirty patients will receive Integrated Neuromuscular Inhibition Technique and mulligan therapy three times a weeks for six weeks+postural correction exercises
  Interventions: Other: Integrated Neuromuscular Inhibition Technique and mulligan therapy; Other: postural correction exercises
- Integrated Neuromuscular Inhibition Technique (Experimental): thirty patients will receive Integrated Neuromuscular Inhibition Technique+postural correction exercises three times a weeks for six weeks
  Interventions: Other: Integrated Neuromuscular Inhibition Technique; Other: postural correction exercises
- mulligan therapy (Experimental): thirty patients will receive mulligan Technique+postural correction exercises three times a weeks for six weeks
  Interventions: Other: mulligan therapy; Other: postural correction exercises
- postural correction exercises (Active Comparator): thirty patients will receive postural correction exercises three times a weeks for six weeks
  Interventions: Other: postural correction exercises

INTERVENTIONS:
Other: Integrated Neuromuscular Inhibition Technique and mulligan therapy — patients will receive Integrated Neuromuscular Inhibition Technique in the form of intermittent ischemic compression, strain counter strain and muscle energy technique and mulligan therapy for limited cervical range of motion
  Arms: Integrated Neuromuscular Inhibition Technique and mulligan therapy
Other: Integrated Neuromuscular Inhibition Technique — patients will receive Integrated Neuromuscular Inhibition Technique in the form of intermittent ischemic compression, strain counter strain and muscle energy technique
  Arms: Integrated Neuromuscular Inhibition Technique
Other: mulligan therapy — patients will receive mulligan therapy for limited cervical range of motion
  Arms: mulligan therapy
Other: postural correction exercises — the patients will receive two strengthening exercises (deep cervical flexors and scapular retractors) and two stretching: cervical extensors (sub-occipital muscles) and pectoral muscles). The program was based on a program by Harman and Kendall

SUMMARY:
this study will be conducted to investigate the impact of adding integrated neuromuscular inhibition technique to mulligan therapy in symptomatic forward head posture.

DETAILED DESCRIPTION:
Forward head posture is anterior positioning of the cervical spine, which is regarded as a "bad" head posture and is commonly found in patients who experience problems with the head and neck. Particularly, forward head posture is frequently found in people sitting in front of a computer for prolonged periods. Load increases in the muscles and joints of the cervical spine as a result of forward head posture are considered a major cause of musculoskeletal disorders. INIT is effective as it causes sustained or intermittent compression which causes ischemia reduces local circulation until pressure is released, after which a flushing of fresh oxygenated blood occurs. Mechanoreceptors impulses interface with slower pain messages reducing amount of pain messges reaching the brain, releasing pain relieving hormones, decreasing myofascial pain. Stretches the taut bands of muscles fibers. INIT along with strengthening excercises proved to be beneficial in decreasing disability improving Range of motion. The concept of SNAG is to increase the treatment effects by having patients perform active movements while removing pain in the lesions by means of manipulative therapy. This is a new concept in the manipulative therapy field, and differs from traditional manipulative therapy by combining the active movements of the patients with additional passive movements performed with the aid of therapists

ELIGIBILITY:
Inclusion Criteria:

* CVA equal or less than 50
* Had cervical pain for more than three months and had visited an orthopedist clinic

Exclusion Criteria:

* cervical spine spondylosis
* fractures or cervical spinal surgery
* Cervical or shoulder neurological movement disorder.
* Temporo-mandibular surgery, (5) Pathologic trauma

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
pain intensity | up to six weeks
  visual analogue scale will be used to asses pain intensity which patient will be instructed to put point on line from no pain to tolerable pain. The scale consists of a line, usually 100 mm long, ranging from no pain or discomfort (zero) , to the worst pain that could possibly feel

SECONDARY OUTCOMES:
neck disability | up to 6 weeks
  will be measured by Arabic neck disability index. It contains ten category/classes. Each category contains six choices (zero-five).Score from zero to four no disability, from five to 15 this is mild, From 15 to 24 this is moderate, from 25 to 34 this is severe, more than 34 this is a complete disability
pressure pain threshold | up to six weeks
  pressure pain threshold pressure pain threshold will be assessed by commander algometer
cervical range of motion | up to six weeks
  range of motion will be measured by inclinometer CROM. The CROM (deluxe version - Performance Attainment Associates, Roseville, MN, USA) measures the cervical range of motion5- for fexion, extension, lateral fexion, and rotation using separate inclinometers. These inclinometers are attached to a frame similar to that for eyeglasses one in the sagittal plane for fexion - extension, second in the frontal plane for lateral fexion and a third in the horizontal plane for rotation.
craniovertebral angle | up to six weeks
  The craniovertebral angle is identified as the intersection of a horizontal line passing through the C7 spinous process and a line joining the midpoint of the tragus of the ear to the skin overlying the C7 spinous process. it measured by photogrametric methods. when the angle less than or equal 50 degree